CLINICAL TRIAL: NCT01006707
Title: fMRI Imaging of Opioid Withdrawal in Healthy Human Volunteers
Brief Title: Functional Magnetic Resonance Imaging of Opioid Withdrawal in Healthy Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Larry Fu-nien Chu, Associate Professor of Anesthesia, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-10212009-4200
Record Dates: First submitted 2009-10-30; First posted 2009-11-03 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron, then Placebo (Other): Some participants received ondansetron pretreatment during the second session, and then placebo during the third session.
  Interventions: Drug: Ondansetron
- Placebo, then Ondansetron (Other): Some participants received placebo pretreatment during the second session, and then ondansetron pretreatment during the third session.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — In this cross-over study, the blinded patient will receive saline placebo in one session and ondansetron in the other. The order is decided with a randomization table. If ondansetron is randomly chosen, an 8mg IV Bolus will be given at the start of the study for 30 minutes by the unblinded investigator.
  Other Names: Zofran

SUMMARY:
Opioid medications are commonly used for pain relief. When given over time, physical dependence can occur. This results in unpleasant side effects--such as agitation and nausea--if opioid medications are suddenly stopped. However, we do not know how withdrawal affects the brain. We know that a medication named Ondansetron can help ease or prevent symptoms associated with opioid withdrawal. Through imaging of the brain by fMRI, we hope to see how opioid withdrawal, with and without the administration of ondansetron, affects brain activity.

DETAILED DESCRIPTION:
During the study, each participant attended three separate lab-based acute opioid withdrawal sessions. The first session was undertaken in a mock MRI scanner and was designed to determine if participants could tolerate withdrawal in the scanning environment. Participants who were able to successfully and safely tolerate opioid withdrawal while in the scanner were approved to continue with the following study sessions. Participants were then pretreated intravenously (IV) with either 0.9% normal saline placebo or 8mg ondansetron. Later, participants in all sessions received IV naloxone (10mg/70kg) to precipitate opioid withdrawal. Participants were assigned to ondansetron or placebo pretreatment conditions in a randomized, double-blinded, and counter-balanced order. Objective Opioid Withdrawal Scale (OOWS) and Subjective Opioid Withdrawal Scale (SOWS) were assessed throughout the study to quantify withdrawal. Study timeline progressed as follows: T=-165, 8mg ondansetron or placebo infusion, T=-135, Morphine infusion (10mg/70kg), T=-41 preparation for MRI, T=-21, start MRI, T=-13, baseline OOWS/SOWS, T=-9, start of fMRI, T=0 Naloxone induced withdrawal, T=5, OOWS, T=15, OOWS, T=20, Retrospective OOWS.

ELIGIBILITY:
Inclusion Criteria

* Patients will be healthy male volunteers, ages 18-35.

Exclusion Criteria

* Females were excluded due to menstrual cycle modulation of opioid response.
* We will exclude individuals with Raynaud's disease or a history of coronary artery disease.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Larry Fu-nien Chu, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Compton P, Miotto K, Elashoff D. Precipitated opioid withdrawal across acute physical dependence induction methods. Pharmacol Biochem Behav. 2004 Feb;77(2):263-8. doi: 10.1016/j.pbb.2003.10.017. PMID 14751453
- [Background] Compton P, Athanasos P, Elashoff D. Withdrawal hyperalgesia after acute opioid physical dependence in nonaddicted humans: a preliminary study. J Pain. 2003 Nov;4(9):511-9. doi: 10.1016/j.jpain.2003.08.003. PMID 14636819
- [Background] Stein EA, Pankiewicz J, Harsch HH, Cho JK, Fuller SA, Hoffmann RG, Hawkins M, Rao SM, Bandettini PA, Bloom AS. Nicotine-induced limbic cortical activation in the human brain: a functional MRI study. Am J Psychiatry. 1998 Aug;155(8):1009-15. doi: 10.1176/ajp.155.8.1009. PMID 9699686
- [Background] Krystal JH, Woods SW, Kosten TR, Rosen MI, Seibyl JP, van Dyck CC, Price LH, Zubal IG, Hoffer PB, Charney DS. Opiate dependence and withdrawal: preliminary assessment using single photon emission computerized tomography (SPECT). Am J Drug Alcohol Abuse. 1995 Feb;21(1):47-63. doi: 10.3109/00952999509095229. PMID 7762544
- [Background] Williams TM, Daglish MR, Lingford-Hughes A, Taylor LG, Hammers A, Brooks DJ, Grasby P, Myles JS, Nutt DJ. Brain opioid receptor binding in early abstinence from opioid dependence: positron emission tomography study. Br J Psychiatry. 2007 Jul;191:63-9. doi: 10.1192/bjp.bp.106.031120. PMID 17602127
- [Background] Hui SC, Sevilla EL, Ogle CW. Prevention by the 5-HT3 receptor antagonist, ondansetron, of morphine-dependence and tolerance in the rat. Br J Pharmacol. 1996 Jun;118(4):1044-50. doi: 10.1111/j.1476-5381.1996.tb15504.x. PMID 8799580
- [Background] Pinelli A, Trivulzio S, Tomasoni L. Effects of ondansetron administration on opioid withdrawal syndrome observed in rats. Eur J Pharmacol. 1997 Dec 11;340(2-3):111-9. doi: 10.1016/s0014-2999(97)01349-6. PMID 9537805
- [Background] Lowe AS, Williams SC, Symms MR, Stolerman IP, Shoaib M. Functional magnetic resonance neuroimaging of drug dependence: naloxone-precipitated morphine withdrawal. Neuroimage. 2002 Oct;17(2):902-10. PMID 12377164
- [Result] Chu LF, Lin JC, Clemenson A, Encisco E, Sun J, Hoang D, Alva H, Erlendson M, Clark JD, Younger JW. Acute opioid withdrawal is associated with increased neural activity in reward-processing centers in healthy men: A functional magnetic resonance imaging study. Drug Alcohol Depend. 2015 Aug 1;153:314-22. doi: 10.1016/j.drugalcdep.2015.04.019. Epub 2015 May 27. PMID 26059463

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Run-in: Participants received pretreatment with placebo to match ondansetron in Study Session 1 prior to randomization to cross-over treatment arms in Study Sessions 2 and 3.
- Ondansetron, Then Placebo: Participants received pretreatment with ondansetron (8mg IV Bolus) in Study Session 2 then placebo to match ondansetron in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
- Placebo, Then Ondansetron: Participants received pretreatment with placebo to match ondansetron in Study Session 2 then ondansetron (8mg IV Bolus) in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
Period: Study Session 1
Arm/Group | Placebo Run-in | Ondansetron, Then Placebo | Placebo, Then Ondansetron
Started | 15 | 0 | 0
Completed (After run-in, participants were randomized to Ondansetron then Placebo, or Placebo then Ondansetron) | 10 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Could not tolerate withdrawal in scanner | 3 | 0 | 0
Period: Study Session 2
Arm/Group | Placebo Run-in | Ondansetron, Then Placebo | Placebo, Then Ondansetron
Started | 0 | 4 | 6
Completed | 0 | 4 | 6
Not Completed | 0 | 0 | 0
Period: Study Session 3
Arm/Group | Placebo Run-in | Ondansetron, Then Placebo | Placebo, Then Ondansetron
Started | 0 | 4 | 6
Completed | 0 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants received placebo during Study Session 1 (placebo run-in), then were randomized to receive pretreatment with ondansetron (8mg IV Bolus) in Study Session 2 then placebo to match ondansetron in Study Session 3, or pretreatment with placebo to match ondansetron in Study Session 2 then ondansetron (8mg IV Bolus) in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10
Weight [Mean (Standard Deviation); unit: kilograms] | 74.33 (4.4)
Height [Mean (Standard Deviation); unit: centimeters] | 177.9 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Brain Regions With Increases or Decreases in Amplitude of Low Frequency Fluctuations (ALFF) Associated With Ondansetron Administration
Description: Changes are reporting using Spearman's correlation coefficient, using within-subject factors of time (pre-naloxone, post-naloxone) and pre-treatment (placebo, ondansetron). Changes in Objective Opioid Withdrawal Scale (OOWS) and Subjective Opioid Withdrawal Scale (SOWS) with correlation coefficient >0.45 are reported. The OOWS consists of 13 observable physical symptoms assessed over a 5-minute observation period and scored as present (score of 1) or absent (score of 0). The total OOWS scores is determined by summing the scores of the 13 items. OOWS scores can range from 0 to 13; lower scores correspond to fewer symptoms. SOWS consists of 16 physical and emotional symptoms rated by the participant on a scale from 0 (not at all) to 4 (extremely), to indicate the extent to which the symptom describes how they are feeling at the time. The total SOWS score is determined by summing the scores of the 16 items. Scores range from 0 to 64; lower scores correspond to fewer symptoms.
Time Frame: 36 minutes
Measure: Number; unit: correlation coefficient
Groups:
- All Ondansetron: All participants received pretreatment with ondansetron (8mg IV Bolus) and with placebo to match ondansetron. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
Arm/Group | All Ondansetron
Number analyzed (Participants) | 10
correlation coefficient
  Left inferior frontal gyrus, orbital (OOWS) | 0.519
  Right inferior frontal gyrus, orbital (OOWS) | 0.562
  Right superior frontal gyrus, medial (SOWS) | 0.478
  Right inferior frontal gyrus, orbital (SOWS) | 0.486
  Left superior temporal gyrus (OOWS) | -0.612
  Left caudate head (SOWS) | 0.475

2. Secondary Outcome: Objective Opioid Withdrawal Scale Score 5 Minutes Following Ondansetron or Placebo Administration
Description: The OOWS consists of 13 observable physical symptoms that are assessed over a five-minute observation period and scored as present (score of 1) or absent (score of 0). The total OOWS scores is determined by summing the scores of the 13 items. OOWS scores can range from a low of 0 to a high of 13. A score of 0 would suggest that no objective signs of withdrawal were observed while a score of 13 would suggest that every observable sign of withdrawal was observed.
Time Frame: 5 Minutes Following Ondansetron or Placebo Administration
Population: Participants completing the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ondansetron: Participants received pretreatment with ondansetron (8mg IV Bolus) in Study Session 2 then placebo to match ondansetron in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
- Placebo: Participants received pretreatment with placebo to match ondansetron in Study Session 2 then ondansetron (8mg IV Bolus) in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 1 (0.5) | 2 (1.3)
Statistical Analysis 1: Comparison: Ondansetron vs Placebo; Results were considered significant at p<0.05; Test type: Superiority or Other; p = 0.042, ANOVA

3. Secondary Outcome: Objective Opioid Withdrawal Scale Score 15 Minutes Following Ondansetron or Placebo Administration
Description: as for outcome 2
Time Frame: 15 Minutes Following Ondansetron or Placebo Administration
Population: Participants completing the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Participants received pretreatment with placebo to match ondansetron in Study Session 2 then ondansetron (8mg IV Bolus) in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 2.7 (1.1) | 2.2 (1.1)
Statistical Analysis 1: Comparison: Ondansetron vs Placebo; Results were considered significant at p<0.05; Test type: Superiority or Other; p = 0.322, ANOVA

4. Secondary Outcome: Subjective Opioid Withdrawal Scale (SOWS) Score 20 Minutes Following Ondansetron or Placebo Administration
Description: The SOWS consists of 16 physical and emotional symptoms that are rated by the participant on a scale from 0 (not at all) to 4 (extremely), to indicate the extent to which the symptom describes how they are feeling at the time. The total SOWS score is determined by summing the scores of the 16 items. Scores range from a low of 0 to a high of 64. A score of 0 would suggest that the individual is experiencing no symptoms of withdrawal while a score of 64 would suggest that the individual is experiencing all 16 symptoms of withdrawal to the fullest extent possible.
Time Frame: 20 minutes following Ondansetron or Placebo administration
Population: Participants completing the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 5.7 (4.5) | 8.1 (7.2)
Statistical Analysis 1: Comparison: Ondansetron vs Placebo; Results were considered significant at p<0.05; Test type: Superiority or Other; p = 0.261, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events data was collected across all study sessions (total of 3 weeks).
Groups:
- Ondansetron: Participants received placebo during Study Session 1 (placebo run-in), then received pretreatment with ondansetron (8mg IV Bolus) in Study Session 2 then placebo to match ondansetron in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
- Placebo: Participants received placebo during Study Session 1 (placebo run-in), then received pretreatment with placebo to match ondansetron in Study Session 2 then ondansetron (8mg IV Bolus) in Study Session 3. Bolus was be given at the start of the study for 30 minutes by the unblinded investigator.
Arm/Group | Ondansetron | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Opioid withdrawal model not necessarily generalizable to individuals with chronic pain and chronic opioid usage; short duration of scan; potential physiological noise in data; unable to obtain strong assessments of OOWS and SOWS during the scan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No